CLINICAL TRIAL: NCT03685396
Title: Patient Morbidity After Palatal Free Gingival Grafts With or Without PRF Membranes Coverage: a Comparative Randomized Clinical Trial
Brief Title: Patient Morbidity After Palatal Free Gingival Grafts With or Without PRF Membranes Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera San Paolo (Other)
Responsible Party: Principal Investigator, Eliam Scaramuzza, Principal investigator, Azienda Ospedaliera San Paolo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRF
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Postoperative Pain; Postoperative Complications; Gingival Recession
Keywords: Connective tissue graft; Platelet concentrates; PRF; Mucogingival surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Gingival Recession | interventions — Hemostasis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): In the Test Group venous blood sampling was done in order to prepare PRF membranes used to cover the donor site of the connective tissue graft.
  Interventions: Biological: Platelet rich fibrin ( PRF)
- Control Group (Active Comparator): In Control Group hemostatic agents with oxidized and regenerated cellulosa were used to cover the donor site.
  Interventions: Drug: hemostatic agents with oxidized and regenerated cellulosa

INTERVENTIONS:
Biological: Platelet rich fibrin ( PRF) — Venous blood was collected with a butterfly needle in two 10 mL tubes without anticoagulants or other chemicals. The tubes were immediately centrifuged at 3000 rpm for 10 minutes.
  At the end of centrifugation a fibrin clot (PRF) was obtained in the middle of the tube, just between the red corpuscles at the bottom and acellular plasma at the top. The PRF clot was taken from the tube and the red cells portion at the base of the clot was eliminated with sterile scissors Then the PRF was enveloped in sterile gauzes and positioned between two glass plates: the compression drove out the serum from the clot obtaining PRF membranes that were ready to be used in the surgical site.
  Arms: Test Group
Drug: hemostatic agents with oxidized and regenerated cellulosa — In the Control Group hemostatic agents with oxidized and regenerated cellulosa were sutured to the palatal wound with mattress suture ( silk 5/0).
  Arms: Control Group

SUMMARY:
This study evaluates postoperative morbidity of patients that undergo free gingival graft harvesting from palate with or without use of autogenous PRF (Platelet Rich Fibrin) membranes to cover the donor site.In the Test Group venous blood sampling was done in order to prepare PRF membranes used to cover the donor site, whereas in Control Group hemostatic agents with oxidized and regenerated cellulosa were used.

ELIGIBILITY:
Inclusion Criteria:

* FMPS (Full Mouth Plaque Score) and FMBS (Full Mouth Bleeding Score) < 20%,
* presence of two adjacent Miller's Class I and II recession defects on natural teeth (≥ 2mm in depth);

Exclusion Criteria:

* contraindications for periodontal surgery
* taking medications or having diseases known to interfere with periodontal tissue health or healing and coagulation.
* smoking more than 10 cigarettes a day
* Gingival recessions on molar teeth were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera San Paolo - Polo Universitario - Università degli Studi di Milano, Milan, Milano, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 subjects were selected from those seeking care at the Department of oral surgery, Dental clinic G.Vogel, San Paolo hospital,Milan.
Groups:
- Test Group: In the Test Group venous blood sampling was done in order to prepare PRF membranes used to cover the donor site of the connective tissue graft.
  Platelet rich fibrin ( PRF): Venous blood was collected with a butterfly needle in two 10 mL tubes without anticoagulants or other chemicals. The tubes were immediately centrifuged at 3000 rpm for 10 minutes.
  At the end of centrifugation a fibrin clot (PRF) was obtained in the middle of the tube, just between the red corpuscles at the bottom and acellular plasma at the top. The PRF clot was taken from the tube and the red cells portion at the base of the clot was eliminated with sterile scissors Then the PRF was enveloped in sterile gauzes and positioned between two glass plates: the compression drove out the serum from the clot obtaining PRF membranes that were ready to be used in the surgical site.
Period: Overall Study
Arm/Group | Test Group | Control Group
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Group | Control Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (6) | 38.4 (5) | 36.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 12 | 6 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain: VAS
Description: The patient morbidity was evaluated with a questionnaire given to patients 1 week following surgery considering parameters such as post-operative pain, discomfort, bleeding, stress and inability to chew. The questionnaire included the evaluation of the intensity of these parameters on a Visual Analogical Scale (VAS) of 100 mm. Patients had to show their level of pain by indicating a position along a continuous line of 100mm between two end-points. The 0 end-point corresponded to abscence of pain, whereas the end-point at 100mm corresponded to the worst level of pain felt in life. Then the point indicated by the patient was measured in millimeters.
Time Frame: 2 weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 21 | 21
score on a scale | 20.00 [12 to 29] | 62 [33 to 80]

2. Primary Outcome: Post-operative Discomfort
Description: Discomfort was defined as the level of soreness experienced by the patients during the first post-operative week due to the palatal wound and how it influenced the ability to work and the quality of the sleep. The questionnaire included the evaluation of the intensity of post-operative discomfort on a Visual Analogical Scale (VAS) of 100 mm. Patients had to show their level of discomfort by indicating a position along a continuous line of 100mm between two end-points. The 0 end-point corresponded to abscence of discomfort whereas the end-point at 100mm corresponded to the worst possible discomfort . Then the point indicated by the patient was measured in millimeters.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 21 | 21
score on a scale | 39 [21 to 40] | 60 [59 to 80]

3. Primary Outcome: Post-operative Stress
Description: Stress was related to the level of apprehension and fear experienced by the patients of jeopardizing the palatal wound. The questionnaire included the evaluation of the intensity of post-operative stress on a Visual Analogical Scale (VAS) of 100 mm. Patients had to show their level of stress by indicating a position along a continuous line of 100mm between two end-points. The 0 end-point corresponded to abscence of stress whereas the end-point at 100mm corresponded to the worst possible stress . Then the point indicated by the patient was measured in millimeters.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 21 | 21
score on a scale | 21 [10 to 49.9] | 50 [29 to 62]

4. Primary Outcome: Post-operative Inability to Chew
Description: Inability to chew was described as the level of variation of the patients' eating habits due to the presence of the palatal wound.
  The questionnaire included the evaluation of the intensity of post-operative inability to chew on a Visual Analogical Scale (VAS) of 100 mm. Patients had to show their level of inability to chew by indicating a position along a continuous line of 100mm between two end-points. The 0 end-point corresponded to abscence of changes in their eating habits whereas the end-point at 100mm corresponded to the worst possible inability to chew. Then the point indicated by the patient was measured in millimeters.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 21 | 21
score on a scale | 60 [39 to 70] | 60 [59 to 80]

ADVERSE EVENTS:
Time Frame: 90 days after surgery
Arm/Group | Test Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03685396/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03685396/SAP_002.pdf